CLINICAL TRIAL: NCT07205341
Title: A Pilot Clinical Study to Assess Correlation Between Arterial Blood Volume Status and Cardiac Efficiency, and HemoCept Device Data in Trans-Aortic Valve Replacement (TAVR} Surgery
Brief Title: Detecting Changes in Arterial Blood Volume and Cardiac Efficiency
Status: Recruiting | Type: Observational
Sponsor: HemoCept Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: PRT-012
Record Dates: First submitted 2025-09-16; First posted 2025-10-03 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-12

CONDITIONS: Aortic Valve Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of this Pilot Study is to demonstrate the efficacy of the Hemocept device in detecting changes in arterial blood volume and cardiac efficiency.

ELIGIBILITY:
Inclusion Criteria:

* Subjects or representatives must have voluntarily signed the informed consent form before any study related procedures.
* Subjects can be any gender but must be between (and including) the ages of 18 and 80.
* Subject ls being treated by the participating healthcare facility .

  ., Subject requires a trans-aortic valve replacement.
* Subject is able and willing to provide informed consent and HIPM authorization.
* Subject is able and willing to meet all study requirements.

Exclusion Criteria:

* Subject is pregnant, breast-feeding, or intends to become pregnant during the course of the study.
* Subject has a personal medical history that includes:

  * Long O-T syndrome
  * Cardiac channelopathies
  * Seizures

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be between 18 and 80 and above who meet all the Inclusion/Exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-04-29 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Correlation of HemoCept device measurements with aortic valve pressure gradient changes. | Perioperative; immediately before procedure, and up to 24 hours after the procedure
  The primary endpoint is the ability of the HemoCept device to properly detect changes consistent with aortic valve pressure gradient values, measured by echocardiogram pre and post TAVR procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Jamie Doucet, MD, Principal Investigator — Boulder Heart
Locations (1):
- Boulder Heart, Boulder, Colorado, United States

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available